CLINICAL TRIAL: NCT00443196
Title: Application of the Microculture Kinetic (MiCK) Assay for Apoptosis to Testing Drug Sensitivity of Ovarian, Fallopian and Primary Peritoneal Adenocarcinomas
Brief Title: Testing Drug Sensitivity of Ovarian, Fallopian and Primary Peritoneal Adenocarcinomas
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pierian Biosciences (Industry)
Responsible Party: Cary Presant, MD, DiaTech Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB 20060042; NCT00531388 (obsolete NCT alias)
Record Dates: First submitted 2006-06-14; First posted 2007-03-05 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2011-03

CONDITIONS: Adenocarcinoma; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Chemosensitivity; Ovarian Cancer; Chemotherapy; Fallopian Adenocarcinoma; Peritoneal Adenocarcinoma; Patients with pathological diagnoses of ovarian, fallopian and primary peritoneal adenocarcinomas.; Patients with de novo malignancies and no previous chemotherapy; Patients with advanced refractory malignancies who received no more than 2 standard chemotherapy treatment protocols.
MeSH Terms: conditions — Adenocarcinoma; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms

ARMS (1):
- Experimental (Experimental)
  Interventions: Procedure: MiCK Assay

INTERVENTIONS:
Procedure: MiCK Assay — Physician determined treatment

SUMMARY:
2.0 Study Objectives: 2.1 To evaluate the ability of the MiCK assay to predict the outcome of chemotherapy of cancer patients for first-line treatment.

2.2 To evaluate the ability of the MiCK assay to guide chemotherapy of cancer patients in a third-line, refractory treatment setting (exclusive of anti-VEGF)

DETAILED DESCRIPTION:
1. 0 Background and Rationale: Despite the use of aggressive treatment protocols, less than 10% of cancer patients with an advanced disease respond to the therapy. There is a variety of different cancer drug regimens, all of which have approximately the same probability of clinical effectiveness. Identification of those patients who will or will not respond to a specific chemotherapy is important for making decisions regarding chemotherapy regimens as well as alternative management approaches. A laboratory test that could help to determine the sensitivity of an individual patient's tumor cells to specific chemotherapeutic agents would be valuable in choosing the optimal chemotherapy regimen for that patient with an expectation of increasing the response rate to the therapy. Several types of in vitro assays that measure tumor cell survival following exposure to cytotoxic agents have been evaluated for their ability to predict chemotherapy outcomes. As a group, these assays are referred to as drug resistance assays. In a resistance assay, the surviving tumor cells can be detected directly by their exclusion or metabolism of specific dyes. Alternatively, since some of tumor cells are proliferating, their survival can be detected by measurement of DNA synthesis by radiolabeled precursor incorporation or demonstration of clonogenic potential by growth into colonies in semi-solid culture medium. In several clinical studies, these assays were useful in detecting drug resistance and in predicting a poor prognosis for cancer patients. However, these resistance assays cannot detect sensitivity of an individual patient's tumor cells to a specific drug. Therefore, new methods determining drug-sensitivity of the tumor cells of an individual patient and, thus, capable of both predicting a positive treatment outcome and guiding chemotherapy, would be of significant value.

Recently, Dr. Kravtsov has developed an automated microculture kinetic (MiCK) assay for measuring drug induced apoptosis in tumor cells. Apoptosis is a distinct mode of cell death which occurs under physiological conditions and yet can be induced in malignant cells by chemical and physical factors including antitumor drugs. During the last decade, it has been recognized that chemotherapeutic agents exert their antitumor activity by triggering apoptosis in susceptible tumor cells. This implies that the MiCK assay for apoptosis provides a mechanism-based approach to studying effects of cytotoxic agents on tumor cells. Unlike "resistance" assays that measure a fraction of cells surviving drug exposure, the MiCK assay measures a fraction of tumor cells killed by a chemotherapeutic agent via mechanism of apoptosis. Therefore the MiCK assay determines drug sensitivity, rather than resistance. Recently the MiCK assay has been shown to predict complete remission rate and survival in acute myeloid leukemia patients better than clinical criteria did. In a limited study, the MiCK assay has been used to direct chemotherapy of the leukemia patients .

The MiCK assay has also been used to study drug-induced apoptosis in solid tumors, including neuroblastoma and colon adenocarcinoma cell lines. More recent data accumulated by DiaTech has demonstrated that the MiCK assay can detect drug induced apoptosis in primary cultures of tumor cells isolated from patients with ovarian carcinoma, gastric carcinoma, metastatic breast cancer and high grade soft tissue sarcoma. Based on these data, we suggest that the MiCK assay may be used to detect drug sensitivity profiles of individual patients with various types of solid tumors. This, in turn, may provide a way to tailor chemotherapy to an individual patient's drug sensitivity profile, and, thus, improve treatment outcomes, decrease adverse effects of the chemotherapy, increase the quality of patient's life, and reduce the treatment cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnoses of ovarian, fallopian and primary peritoneal adenocarcinomas.
* Patients with de novo malignancies and no previous chemotherapy
* Patients with advanced refractory malignancies who received no more than 2 standard chemotherapy treatment protocols.
* Patients of any age group.
* Patients must have tumor which is accessible and agree to undergo biopsies, or drainage of effusions.
* Patients for whom chemotherapy is a treatment option.
* Explanations: We anticipate that newly diagnosed patients will be mostly used to evaluate the ability of the MiCK assay to predict the outcome of the chemotherapy (Objective #2.1) and to establish criteria correlating numerical response in the MiCK assay with probability of the clinically established complete remission. The patients with refractory malignancies will be mostly used to evaluate the ability of the MiCK assay to guide cancer chemotherapy (Objective #2.2). Patients will be seen and managed as outpatients or inpatients, depending on a clinical standard of the institution

Exclusion Criteria:

* Patients with symptomatic/uncontrolled parenchimal brain metastasis and not accessible tumors.
* Patients with meningeal metastasis.
* Patients for whom chemotherapy clinically is not indicated.
* Pregnancy. During the course of the study, all patients of childbearing potential should be instructed to contact the treating physician if they suspect they might have conceived a child; for females, a missing or late menstrual period should be reported to the treating physician. If pregnancy is confirmed by a pregnancy test, the patient must not receive study medication and must not be enrolled into the study or, if already enrolled, must be withdrawn from the study. If a male patient is suspected of having fathered a child while on the study drugs, the pregnant female partner must be notified and counseled regarding the risk to the fetus. Pregnancy during the course of this study will be reported to the Principal Investigator as a serious adverse event. Women of child bearing potential are defined to include any female who has experienced menarche and has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal (defined as amenorrhea for more than 12 consecutive months); these includes also females using oral, implanted, or injectable contraceptive hormones, mechanical devices, or barrier methods to prevent pregnancy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-03; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Complete Response, No Response | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Cary Presant, MD, Principal Investigator — Pierian Biosciences
Locations (1):
- Southeastern Gynecologic Oncology, Atlanta, Georgia, United States